CLINICAL TRIAL: NCT05924737
Title: Delta Waves and Cognitive Recovery During a Restricted Sleep Opportunity After Total Sleep
Brief Title: Delta Waves and Cognitive Recovery
Acronym: RECOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Collaborators: Hotel Dieu de France Hospital (Other); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023_RECOPS; 2023-A01221-44 (Other: IDRCB)
Record Dates: First submitted 2023-06-12; First posted 2023-06-29 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Sleep Deprivation; Cognitive Impairment
Keywords: recovery; sleep
MeSH Terms: conditions — Sleep Deprivation; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Sleep deprivation followed by a short and a long recovery nigjht
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep (Experimental): Sleep deprivation
  Interventions: Other: Sleep deprivatin; Other: Sleep recovery

INTERVENTIONS:
Other: Sleep deprivatin — 40 hours of continuous awakening
Other: Sleep recovery — sleep recovery after 40 hours of continuous awakening

SUMMARY:
In a laboratory protocol in healthy adults, exposed to a prolonged period of wakefulness with a restricted opportunity for sleep (40h of wakefulness / 3h of sleep / 21h of wakefulness), we hypothesize that the relative increase in spectral power of Delta waves [ 1 - 4 Hz] in NREM in the frontal territory, identified as a potential marker of the restorative function of sleep, during a night of sleep with limited recovery (3 h of time in bed) after sleep deprivation (40 h of continuous wakefulness), will be less important in subjects with poor recovery in terms of cognitive performance than in those with good recovery.

DETAILED DESCRIPTION:
Exposure to sleep debt is one of the many stresses to which military personnel are exposed, during operational deployments or high-intensity training1.

The kinetics of cognitive performance degradation during acute sleep restriction or deprivation are relatively well studied in the literature2, with significant inter-individual variability. Restoring these cognitive functions requires sufficient sleep, sometimes for several days. However, the military work environment often offers only limited opportunities for recovery, which does not allow for ad integrum restoration of cognitive capacities, although some subjects recover better than others.

This is problematic in an environment where individual and collective performance levels are a prerequisite for safety and mission success3.

In this context, early identification of poor recuperators, who do not sufficiently restore their cognitive performance after periods of rest, would enable us to adapt more effectively the use of different countermeasures (sleep extension, naps, adapted use of caffeine...)4. This implies the availability of validated objective markers, as subjective assessments are often inadequate in this context. The temporal data classically derived from the analysis of sleep macrostructure (total sleep time, duration of wakefulness after falling asleep, time spent in the various sleep stages, etc.) are compromised when the opportunity for sleep is restricted. It therefore becomes pertinent to look for non-temporal markers that would testify to the efficiency of sleep's recuperative function.

Delta slow waves [1 - 4 Hz], which are mainly observed during deep slow-wave sleep on a sleep EEG, appear to be one of the indicators of the restorative function of sleep. They have been identified as a marker of sleep pressure5. The spectral power in this frequency range (delta power or slow-waves activity), obtained after fast Fourier transformation, bears witness to the activity of these waves. It is known to increase at the start of the night, particularly after sleep debt, and then gradually decrease, reflecting the dissipation of sleep pressure. It is recognized that high spectral power in this frequency range, particularly in deep slow wave sleep, is a marker of the "depth" of sleep" . This depth could guarantee the restorative function of sleep. [...]

In a laboratory protocol in healthy adults, exposed to a prolonged period of wakefulness with a restricted opportunity for sleep (40h of wakefulness / 3h of sleep / 21h of wakefulness), we hypothesize that the relative increase in spectral power of Delta waves [ 1 - 4 Hz] in NREM in the frontal territory, identified as a potential marker of the restorative function of sleep, during a night of sleep with limited recovery (3 h of time in bed) after sleep deprivation (40 h of continuous wakefulness), will be less important in subjects with poor recovery in terms of cognitive performance than in those with good recovery.

ELIGIBILITY:
Inclusion Criteria

* Healthy volunteer man or woman
* Between 18 and 45 years of age
* Having given written consent after having been informed of the terms of the study and the objectives of the genetic analysis performed

Exclusion Criteria:

* Current medical treatment
* Chronic medical pathology, (psychol, cardiovascular or respiratory, sleep disorders)
* Pregnancy
* Sleep disorder
* Extreme chronotype
* Excessive daytime sleepiness
* Suspicion of anxiety or depressive disorder
* Estimated caffeine consumption > 200mg/day
* Not covered by a health insurance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Delta power | One night
  EEG Delta power in Hz

SECONDARY OUTCOMES:
Cognitive performance | 2 days
  Performance during PVT Test, in ms

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de recherche biomédical des armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: No